CLINICAL TRIAL: NCT03947060
Title: BI-SENSES: Validation of Nasal Versus Frontal Placement of the SedLine® Sensor Through Processed Electroencephalography in Adult Patients Undergoing General Anesthesia
Brief Title: The Alternative Position for the SedLine® Sensor
Status: Completed | Type: Observational
Sponsor: Cleveland Clinic Abu Dhabi (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Boris Tufegdzic, Asst Prof Dr Boris Tufegdzic, Cleveland Clinic Abu Dhabi
Other Study IDs: A-2019-028
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Depth of Anesthesia Monitoring
Keywords: Depth of anesthesia; SedLine® sensor; Alternative position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasal & Frontal sensor position: One group of participants with two modes of measurement. First mode is standard frontal placement of the SedLine® sensor. Second mode is alternative nasal placement of the SedLine® sensor.

SUMMARY:
SedLine® Brain Function Monitoring provides real-time insight into a patient's depth of anesthesia with bilateral data acquisition and processing of electroencephalogram (EEG) signals. Four active EEG leads collect data from the frontal lobe with a sensor position on the patient's forehead.

Whenever a frontal approach for neurosurgical procedures is required or the frontal placement of the EEG is not indicated, it would not be possible to place the SedLine® .

Numerous studies have analyzed the change of position and the application of alternative positions for other devices used in assessing the depth of anesthesia. Albeit, yet to date, there is no study that analyzed the application of alternative positions for the SedLine® sensor.

DETAILED DESCRIPTION:
The purpose of study is to compare the standard forehead placement versus a nasal placement of SedLine® sensor for neuromonitoring.

The hypothesis is that placing the central sensors in the montage approximately 2 cm below the standard recommended placement, across the nasal bridge and then running under the eyes to the normal temporal leads placement would put the entire montage out of the operative field and would still have corresponding values and EEG signals.

The primary outcome measure is to monitor and compare processed electroencephalograph (EEG) values (PSi- Patient State Index, SEFL- Spectral Edge Frequency Left, SEFR- Spectral Edge Frequency Right, SR-Suppression Ratio, EMG-Electromyography, ARTF-Artifact) and EEG waveforms, on both sensors (standard-Forehead and alternative-Nasal)

Other parameters that will be measure are patient demographics (age, sex, surgery, ASA status, weight, height, BMI).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age, both genders.
* Patients undergoing simple or complex surgery.
* American Society of Anesthesiologists Classification (ASA) score I to III.

Exclusion Criteria:

American Society of Anesthesiologists Classification (ASA) score IV and V.

* Emergency cases
* Cognitive/Mentally impaired or unable to provide consent
* Previous neurological problems affecting EEG
* Dementia
* Use of sedative or drugs that can alter EEG readings
* Patients under head and neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For each of the two modes of measurement, 1800 data points per subject (1 reading every 2 seconds for 1 hour) per hour will be collected. Assuming a maximum interclass correlation coefficient of .90, a sample size of 40 patients will be required to test the null hypotheses that the two modes of measurement share 95% of their variance via the construction of a 95% confidence interval that ranges no more than +/-5%.
  Data from the 2 placements will be compared and analyzed using a Bland-Altman analysis, a Scatter plot analysis, and a matched-pair analysis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Validation of nasal SedLine® EEG sensor position for monitoring the depth of anesthesia using processed electroencephalograph values | One year
  Determine whether it is possible to apply an alternative SedLine® EEG sensor position in a situation where a standard-forehead position is not possible.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Tufegdzic, MD, Principal Investigator — Cleveland Clinic Abu Dhabi
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03947060/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03947060/ICF_001.pdf